CLINICAL TRIAL: NCT02170376
Title: The Effect of BIA 9-1067 at Steady-state on the Levodopa Pharmacokinetics When Administered With Immediate-release 100/25 mg Levodopa/Carbidopa in Healthy Subjects
Brief Title: The Effect of BIA 9-1067 at Steady-state on the Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-91067-124
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); BIA 9-1067; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Placebo once-daily for 11 days 200 mg entacapone concomitantly with levodopa/carbidopa on Day 12
  Interventions: Drug: Entacapone; Drug: Placebo; Drug: Levodopa/carbidopa
- Group 2 (Experimental): 25 mg BIA 9-1067 once-daily for 11 days Placebo concomitantly with levodopa/carbidopa on Day 12
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/carbidopa
- Group 3 (Experimental): 50 mg 9-1067 once-daily for 11 days Placebo concomitantly with levodopa/carbidopa on Day 12
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/carbidopa
- Group 4 (Experimental): 75 mg 9-1067 once-daily for 11 days placebo concomitantly with levodopa/carbidopa on Day 12
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/carbidopa
- Group 5 (Placebo Comparator): placebo once-daily for 11 days placebo concomitantly with levodopa/carbidopa on Day 12
  Interventions: Drug: Placebo; Drug: Levodopa/carbidopa

INTERVENTIONS:
Drug: BIA 9-1067 — BIA 9-1067 25 mg and 50 mg
  Other Names: Opicapone, OPC
  Arms: Group 2; Group 3; Group 4
Drug: Entacapone — Entacapone (ENT), over-encapsulated tablet 200 mg
  Other Names: Comtan®, ENT
  Arms: Group 1
Drug: Placebo — PLC, placebo
  Other Names: PLC, placebo
Drug: Levodopa/carbidopa — Levodopa/carbidopa, tablet 100/25 mg
  Other Names: Sinemet®

SUMMARY:
The purpose of this study is to determine the effect of repeated dosing of once-daily 25, 50 and 75 mg opicapone (OPC, development code BIA 9-1067) on the levodopa pharmacokinetics (PK), in comparison to placebo and 200 mg entacapone (ENT).

DETAILED DESCRIPTION:
This study was a single-centre, randomized, double-blind, gender-balanced, placebo-controlled study in 4 groups of 20 healthy subjects each (10 male and 10 female). The clinical part included a screening examination within 3 weeks before the first institutionalization, an ambulatory period of 11 days (from Day 1 evening to Day 11 evening), during which the subjects returned to the clinical unit every evening, followed by an institutionalization of 1.5 days (from Day 11 evening to Day 13 morning (i.e. 14 h after the third administration of levodopa/carbidopa). Then, a follow-up visit at 5 to 9 days after collection of the last PK blood sample (i.e. Day 13). The maximum total duration of the clinical study, including the 21-day screening period and the post-study follow-up, was expected to be about 39 to 43 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers 18 to 45 years old (inclusive),
* Body Mass Index (BMI) in normal range (18-30 kg/m²),
* Healthy as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, complete neurological examination and 12-lead ECG (electrocardiogram),
* Negative tests for Hepatitis B surface antigen (HBsAG), anti-Hepatitis C virus (HCV) antibodies and Human immunodeficiency virus (HIV) -1 and HIV-2 antibodies at screening,
* Negative screen for drugs of abuse and alcohol at screening and admission to the treatment period,
* If of childbearing potential (i.e. except if they had been sterilized for at least 3 months or postmenopausal for at least one year - the menopause was defined by a follicule stimulating hormone (FSH) level > 30 IU/L): used a non hormonal acceptable contraception method, i.e. intra-uterine device, condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository for all the duration of the study,
* If female of childbearing potential, had a negative human chorionic gonadotropin (HCG) beta serum pregnancy test at screening and urinary pregnancy test at admission to both ambulatory and confinement periods,
* Non-smokers or ex-smokers for at least 3 months,
* Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study,
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form,
* Registered with the French Social Security in agreement with the French law on biomedical experimentation

Exclusion Criteria:

* Did not conform to the above inclusion criteria, or in case of volunteers who had a clinically relevant surgical history, a clinically relevant family history; had a history of relevant atopy,
* Had a significant infection or known inflammatory process at screening or admission to the treatment period; acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to the treatment period,
* Were vegetarians, vegans or had medical dietary restrictions,
* Could not communicate reliably with the Investigator,
* Were unlikely to co-operate with the requirements of the study; history of hypersensitivity to OPC, tolcapone, ENT, levodopa, carbidopa, benserazide or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs,
* Had any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, hematological, neurological, or psychiatric disease,
* Presented any clinically significant illness in the previous 28 days before Day 1 of this study; history of drug abuse within 1 year before study Day 1; history of alcoholism within 1 year before Day 1,
* Had taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the dose administration,
* Consumed more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g,
* Drank more than 8 cups daily of beverage containing caffeine,
* Had poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician,
* Had received any experimental drug within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health,
* Forfeited their freedom by administrative or legal award or were under guardianship,
* Had undergone surgery or had donated blood (i.e. 450 mL) within 12 weeks before study Day 1,
* Had positive urine screening of ethyl alcohol or drugs of abuse upon admission to the treatment period,
* Had any history of tuberculosis and/or prophylaxis for tuberculosis; positive results to HIV, HBsAg or anti-HCV tests; participation in any previous clinical study with OPC,
* If female, was pregnant or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS aster, Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Placebo Then Entacapone/Levodopa: Placebo once-daily for 11 days 200 mg entacapone concomitantly with levodopa/carbidopa on Day 12
  Entacapone: Entacapone (ENT), over-encapsulated tablet 200 mg
  Placebo: PLC, placebo
  Levodopa/carbidopa: Levodopa/carbidopa, tablet 100/25 mg
- Group 2: BIA 25 mg Then Placebo/Levodopa/Carbidopa: 25 mg BIA 9-1067 once-daily for 11 days Placebo concomitantly with levodopa/carbidopa on Day 12
  BIA 9-1067: BIA 9-1067 25 mg and 50 mg
  Placebo: PLC, placebo
  Levodopa/carbidopa: Levodopa/carbidopa, tablet 100/25 mg
- Group 3: BIA 50 mg Then Placebo/Levodopa/Carbidopa: 50 mg 9-1067 once-daily for 11 days Placebo concomitantly with levodopa/carbidopa on Day 12
  BIA 9-1067: BIA 9-1067 25 mg and 50 mg
  Placebo: PLC, placebo
  Levodopa/carbidopa: Levodopa/carbidopa, tablet 100/25 mg
- Group 4: BIA 75 mg Then Placebo/Levodopa/Carbidopa: 75 mg 9-1067 once-daily for 11 days placebo concomitantly with levodopa/carbidopa on Day 12
  BIA 9-1067: BIA 9-1067 25 mg and 50 mg
  Placebo: PLC, placebo
  Levodopa/carbidopa: Levodopa/carbidopa, tablet 100/25 mg
- Group 5: Placebo Then Levodopa/Carbidopa: placebo once-daily for 11 days placebo concomitantly with levodopa/carbidopa on Day 12
  Placebo: PLC, placebo
  Levodopa/carbidopa: Levodopa/carbidopa, tablet 100/25 mg
Period: Overall Study
Arm/Group | Group 1: Placebo Then Entacapone/Levodopa | Group 2: BIA 25 mg Then Placebo/Levodopa/Carbidopa | Group 3: BIA 50 mg Then Placebo/Levodopa/Carbidopa | Group 4: BIA 75 mg Then Placebo/Levodopa/Carbidopa | Group 5: Placebo Then Levodopa/Carbidopa
Started | 16 | 16 | 16 | 16 | 16
Pharmacokinetic Population | 16 | 15 | 16 | 16 | 16
Completed | 16 | 15 | 16 | 16 | 16
Not Completed | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 16 | 16 | 16 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 8 | 8 | 40
  Male | 8 | 8 | 8 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration of Levodopa
Description: Cmax - Maximum plasma concentration of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone.
Time Frame: pre-first dose and at 0.5, 1.0, 1.5, 2.0, 3.0, 4.0 and 5.0 h post-first and -second levodopa/carbidopa administration, and at 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 8.0 and 14.0 h post-third levodopa/carbidopa administration
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- OPC 25 mg: OPC: BIA 9-1067 25 mg
- OPC 50 mg: OPC: BIA 9-1067 50 mg
- OPC 75 mg: OPC: BIA 9-1067 25 mg and 50 mg
- ENT 200 mg: Entacapone (ENT), over-encapsulated tablet 200 mg
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
ng/mL
  Post First Dose | 1047 (340) | 1203 (453) | 1030 (400) | 1057 (335) | 876 (328)
  Post Second Dose | 1550 (542) | 1619 (762) | 1974 (847) | 2113 (868) | 1437 (569)
  Post Third Dose | 1268 (532) | 1393 (627) | 1346 (337) | 1658 (435) | 1303 (518)

2. Primary Outcome: Tmax - Time of Occurrence of Maximum Plasma Concentration
Description: Tmax - Time to Reach maximum plasma concentration of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
hours
  Post First Dose | 1.31 (0.854) | 1.13 (0.790) | 1.34 (1.01) | 1.28 (0.515) | 1.13 (0.695)
  Post Second Dose | 0.875 (0.465) | 1.20 (0.862) | 1.06 (0.892) | 1.19 (0.854) | 0.906 (0.491)
  Post Third Dose | 1.69 (0.964) | 1.33 (0.699) | 1.34 (0.65) | 1.31 (0.854) | 1.59 (0.861)

3. Primary Outcome: AUC0-∞ - Area Under the Concentration-time Curve From Time Zero up to Infinity With Extrapolation of the Terminal Phase
Description: AUC0-∞ of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
ng.h/mL
  Post First Dose | 2305 (391) | 3732 (1418) | 3363 (1042) | 3998 (1275) | 2752 (540)
  Post Second Dose | 3070 (396) | 4967 (2003) | 5727 (1495) | 6213 (1440) | 4367 (1463)
  Post Third Dose | 3299 (433) | 5614 (2467) | 5912 (1478) | 7177 (1835) | 4707 (363)

4. Primary Outcome: AUC0-t - Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Time (t) Corresponding to the Last Quantifiable Concentration.
Description: AUC0-t - of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
ng.h/mL
  Post First Dose | 1985 (346) | 2665 (867) | 2383 (699) | 2829 (794) | 2041 (671)
  Post Second Dose | 2774 (353) | 3678 (1455) | 4151 (1070) | 4597 (1041) | 3445 (1128)
  Post Third Dose | 3123 (447) | 5391 (2444) | 5685 (1466) | 6928 (1797) | 4366 (1426)

5. Primary Outcome: AUC0-5 - AUC Over 5 Hours
Description: AUC0-5 - of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
ng.h/mL
  Post First Dose | 1985 (346) | 2665 (867) | 2383 (699) | 2829 (794) | 2042 (669)
  Post Second Dose | 2774 (353) | 3678 (1455) | 4151 (1070) | 4597 (1041) | 3446 (1125)
  Post Third Dose | 2719 (492) | 3802 (1549) | 3940 (1022) | 4882 (1246) | 3468 (1108)

6. Primary Outcome: t1/2 - Terminal Plasma Half-life
Description: t1/2 - Terminal plasma half-life of levodopa (mean pharmacokinetic parameter) following first oral administration of 100/25 mg levodopa/carbidopa on Day 12 with 25, 50 and 75 mg OPC or placebo and 200 mg Entacapone.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | OPC 25 mg | OPC 50 mg | OPC 75 mg | ENT 200 mg
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Hours
  Post First Dose | 1.46 (0.406) | 2.47 (0.830) | 2.47 (0.098) | 2.39 (0.556) | 2.11 (0.626)
  Post Second Dose | 1.41 (0.136) | 2.23 (0.385) | 2.46 (0.312) | 2.23 (0.513) | 2.09 (0.486)
  Post Third Dose | 1.74 (0.349) | 2.56 (0.440) | 2.75 (0.513) | 2.70 (0.462) | 2.20 (0.632)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 9/16 | 5/16 | 8/16 | 8/16 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=16) | Group 2 (N=16) | Group 3 (N=16) | Group 4 (N=16) | Group 5 (N=16)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 8 | 8 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 5 | 2 | 2 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 2
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pityriasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 3 | 2 | 1
Varicophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other